CLINICAL TRIAL: NCT03566654
Title: A Random Controlled, Double-Blind Clinical Trial: Remote Ischemic Conditioning and Hypertension
Brief Title: Clinical Trial on Remote Ischemic Conditioning and Hypertension（HOPE）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, Professor of Neurosurgery, Vice-President of Xuan Wu Hospital, Capital Medical University, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIC-HP
Record Dates: First submitted 2018-03-27; First posted 2018-06-25 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Essential Hypertension
Keywords: remote ischemic conditioning
MeSH Terms: conditions — Essential Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remote ischemic conditioning (Experimental): Receiving remote ischemic conditioning (RIC) treatment with pressure set at 200 mmHg.
  Interventions: Device: remote ischemic conditioning; Device: ambulatory blood pressure monitoring
- placebo remote ischemic conditioning (Sham Comparator): Receiving sham RIC treatment with pressure set at 50~60 mmHg
  Interventions: Device: ambulatory blood pressure monitoring; Device: Sham remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on unilateral arms and inflated to 200 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeately for 5 times， two times per day. The duration of the treatment is 30+/-2days.
  Other Names: RIC
  Arms: remote ischemic conditioning
Device: ambulatory blood pressure monitoring — A diagnostic technique for measuring blood pressure in daily life by means of automatic intermittent timing. Because ABPM has overcome the limitations of clinic blood pressure measurement, observation error and white coat effect, it can objectively reflect the actual level and fluctuation of blood pressure. Each patient of the two arms will use ABPM measure blood pressure before and after RIC or sham RIC treatment.
  Other Names: ABPM
Device: Sham remote ischemic conditioning — Sham RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on unilateral arms and inflated to 60 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeately for 5 times. The duration of the treatment is 30+/-2days.
  Arms: placebo remote ischemic conditioning

SUMMARY:
Nowadays, the incidence of stroke in China has reached 1.6‰, and this disease has became a primary cause of death in China. One of its major risk factors is hypertension. As shown in the researches, the risk of stroke grows remarkably when the blood pressure increases and there exists a log-linear relationship between them. Systolic pressure and diastolic pressure relate to the risk of stroke independently. Systolic pressure decreasing 10mmHg will reduce the stroke risk by 31% and decrease of 1~3mmHg will reduce the stroke risk by 20~30%. As to diastolic pressure, 5mmHg decrease of it will reduce the stroke risk by 34% and 10mmHg decrease of it will reduce the stroke risk by 56%. In addition, patients with isolated systolic hypertension (SPB≥160mmHg, DPB≤90mmHg) or critical isolated systolic hypertension (SPB=140~159mmHg, DPB< 90mmHg) will suffer a higher risk of stroke than people with normal blood pressure. The ACC has already revised its Hypertension Management Guidelines of standard of diagnosis for hypertension and timing of starting medical treatment in hypertensive patients.Because more and more reseaches shown that people with blood pressure between 120-139/80-89mmHg have higher risk of ASCVSD compared to those with blood pressure lower than 120/80mmHg; However, in China, the diagnostic criteria for hypertension has not been revised yet. Therefore, we still have blind spot in treating such patients who suffer from borderline systolic hypertension at 130~140 mmHg of blood pressure with or without ASCVD or those with the first stage hypertension but refusing to take anti-hypertension drugs. What is more, most of them are middle-aged adults, once they have stroke, it would lead terrible and costly consequences to both their family and the society. Thus, it is necessary to explore new non-pharmacological methods to control blood pressure for reducing the risk of stroke.

DETAILED DESCRIPTION:
There already have had some researchers found the phenomenon of lowing blood pressure among heart failure patients and pre-hypertensive individuals after a long-term of ischemic conditioning therapy. However, there's still lack of specific clinical trials carried out to confirm itspotential treatment effect of lowing blood pressure.

The investigators designed this randomized, doubleblind, controlled clinical trial to examine (1) whether RIC has a beneficial effect on blood pressure; (2) whether RIC exert its protection effect through immunological regulation. There are 2 arms in this trial: One arm is RIC treatment, the other one is sham RIC treatment. Blood pressure will be measured by ambulatory blood pressure monitoring before and after the treatment to evaluate its exact effect on BP. Also, circulatory immunological factors will be tested before and after the treatment to illustate whether immunological regulation involved in the process.

ELIGIBILITY:
Inclusion Criteria:

1. ABPM measures systolic and diastolic blood pressure within the range of 125-145/75-90mmHg;
2. Essential hypertension;
3. without use anti-hypertensive drugs;
4. Written consent was obtained from the subject.

Exclusion Criteria:

1. patients already have had anti-hypertensive drugs;
2. patiets with diabetes mellitus and have a poor blood glucose control;
3. patients with atrial fibrillation or other kinds of arrhythmia;

7. unstable general condition; 8.Subject participating in a study involving other drug or device trial study; 9. patients that investigators think is not suitable.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
changes of blood pressure | 0-33 days
  systolic, diastolic and average blood pressure changes would be tested after interventions by using ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
changes of the circulatory inflammatory factors | 0-33 days
  circulatory inflammatory factors will be tested before and after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD,Ph.D, Principal Investigator — Capital Medical University Xuan Wu Hospital
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes